CLINICAL TRIAL: NCT04656990
Title: SKIPping With PAX: An Integrated Gross Motor and Social-Emotional Skill Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Ali Brian, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00091603
Record Dates: First submitted 2020-11-16; First posted 2020-12-07 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Gross Motor Development Delay; Social Skills; Social Behavior; Sedentary Behavior
MeSH Terms: conditions — Social Skills; Social Behavior; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gross motor and social-emotional integrated intervention group (Experimental): Participants will receive a nine-month intervention which focuses on gross motor skills, physical activity, and social-emotional skills.
  Interventions: Behavioral: Integrated Intervention
- Control (No Intervention): Participants will receive the center's everyday business as usual curriculum.

INTERVENTIONS:
Behavioral: Integrated Intervention — Gross motor and social-emotional integrated intervention
  Arms: Gross motor and social-emotional integrated intervention group

SUMMARY:
The purpose of this study was to test the effects of an integrated intervention on the gross motor and social-emotional development of rural preschool boys and girls. A secondary purpose was to examine intervention effects on physical activity and sedentary behavior. An exploratory aim was to examine the role of executive functioning skills on intervention outcomes. This study featured a repeated measures (baseline, six-month posttest, three month retention [nine-month follow-up]), control group, experimental design. Classrooms were randomly assigned to either the experimental or control groups. Experimental participants received intervention while control participants received business as usual curricula.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the early childhood center, aged 4-5 years

Exclusion Criteria:

* Enrolled in special education classroom

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 277 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lexington 4 Early Childhood Center, Swansea, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: classrooms
Period: Baseline
Arm/Group | Gross Motor and Social-emotional Integrated Intervention Group | Control
Started | 129; 7 classrooms | 148; 7 classrooms
Completed | 109; 7 classrooms | 124; 7 classrooms
Not Completed | 20; 0 classrooms | 24; 0 classrooms
Not completed — pandemic | 20 | 24
Period: Intervention
Arm/Group | Gross Motor and Social-emotional Integrated Intervention Group | Control
Started | 109; 7 classrooms | 124; 7 classrooms
Completed | 109; 7 classrooms | 124; 7 classrooms
Not Completed | 0; 0 classrooms | 0; 0 classrooms
Period: Follow Up Period
Arm/Group | Gross Motor and Social-emotional Integrated Intervention Group | Control
Started | 109; 7 classrooms | 124; 7 classrooms
Completed | 48; 7 classrooms | 51; 7 classrooms
Not Completed | 61; 0 classrooms | 73; 0 classrooms
Not completed — Lost to Follow-up | 61 | 73

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gross Motor and Social-emotional Integrated Intervention Group | Control | Total
Number analyzed (Participants) | 109 | 124 | 233
Age, Continuous [Mean (Standard Deviation); unit: Months] | 60.88 (6.67) | 61.15 (7.14) | 61.03 (6.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 64 | 118
  Male | 55 | 60 | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 15 | 16 | 31
  White | 71 | 83 | 154
  Hispanic | 20 | 20 | 40
  More than one race | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Test of Gross Motor Development, Third Edition
Description: Gross motor development assessment ranges from 0-100 with higher scores reflecting better performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gross Motor and Social-emotional Integrated Intervention Group | Control
Number analyzed (Participants) | 109 | 124
score on a scale | 41.99 (14.40) | 43.36 (13.26)

2. Primary Outcome: Test of Gross Motor Development, Third Edition
Description: Gross motor development assessment ranges from 0-100 with higher scores reflecting better performance.
Time Frame: six-month posttest
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gross Motor and Social-emotional Integrated Intervention Group | Control
Number analyzed (Participants) | 109 | 124
score on a scale | 62.36 (12.35) | 49.75 (11.70)
Statistical Analysis 1: Comparison: Gross Motor and Social-emotional Integrated Intervention Group vs Control; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Slope = 17.10

3. Primary Outcome: Test of Gross Motor Development, Third Edition
Description: Gross motor development assessment ranges from 0-100 with higher scores reflecting better performance.
Time Frame: three-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gross Motor and Social-emotional Integrated Intervention Group | Control
Number analyzed (Participants) | 48 | 51
score on a scale | 51.02 (10.97) | 46.39 (12.05)

4. Primary Outcome: Social Skills Improvement System Rating Scales
Description: Social-Emotional scores range from 0-160 with higher scores reflecting better performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gross Motor and Social-emotional Integrated Intervention Group | Control
Number analyzed (Participants) | 109 | 124
score on a scale | 85.63 (21.65) | 96.38 (20.33)

5. Primary Outcome: Social Skills Improvement System Rating Scales
Description: Social-Emotional scores range from 0-160 with higher scores reflecting better performance.
Time Frame: six-month posttest
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gross Motor and Social-emotional Integrated Intervention Group | Control
Number analyzed (Participants) | 109 | 124
score on a scale | 89.24 (20.30) | 93.03 (21.29)
Statistical Analysis 1: Comparison: Gross Motor and Social-emotional Integrated Intervention Group vs Control; Test type: Superiority; p = 0.04, Mixed Models Analysis; Slope = 3.40

6. Primary Outcome: Social Skills Improvement System Rating Scales
Description: Social-Emotional scores range from 0-160 with higher scores reflecting better performance.
Time Frame: three-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gross Motor and Social-emotional Integrated Intervention Group | Control
Number analyzed (Participants) | 48 | 51
score on a scale | 86.27 (16.77) | 93.00 (22.82)

7. Secondary Outcome: Physical Activity From Accelerometer
Description: The accelerometer, which children wear throughout the day, records step counts which are then converted into numerical representation of levels of physical activity.
Time Frame: Baseline
Population: No data were collected on this measure for the following reason. Because of restrictions emanating from the pandemic, school authorities did not permit children to wear the accelerometers. Consequently, it was not possible to implement this measure. Consequently the number of participants with data on this measure was zero, and the number of participants analyzed on this measure was zero.
Arm/Group | Gross Motor and Social-emotional Integrated Intervention Group | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline, during intervention, posttest, follow up for a total of 12 months
Description: Participants did not partake in any activities that would stray or differ from what could potentially be offered in a school setting.
Arm/Group | Gross Motor and Social-emotional Integrated Intervention Group | Control
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/148
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/148
Other Adverse Events (participants affected / at risk) | 0/129 | 0/148

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT04656990/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT04656990/ICF_001.pdf